CLINICAL TRIAL: NCT01771718
Title: Non-invasive Skin Imaging Using Multiphoton Microscopy
Brief Title: Pilot Study on In-vivo Non-invasive Skin Imaging Using Multiphoton Microscopy
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Kristen Kelly, Professor and Chair, Department of Dermatology, University of California, Irvine
Other Study IDs: 20118494; R01EB026705 (NIH)
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Skin Lesion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Human skin: Multiphoton microscopy imaging to collect information about changes in skin cells and fibrilar structure.
  Interventions: Device: Multiphoton microscopy-based tomograph.

INTERVENTIONS:
Device: Multiphoton microscopy-based tomograph. — non-invasive optical biopsy

SUMMARY:
The purpose of this pilot study is to employ multiphoton microscopy to non-invasively image in-vivo pigmented and non-pigmented human skin lesions for characterization of their morphologic and functional features.

DETAILED DESCRIPTION:
This study is performed using a multiphoton microscopy-based tomograph (MPTflex) developed by JenLab, GmbH (Germany) and a MPM imaging system developed at BLI: Fast Large Area Multiphoton Exoscope (FLAME) to image non-invasively normal and lesional skin. Skin lesions are imaged by multiphoton microscopy and images are compared to those obtained from histopathology through standard of care processed skin biopsies.

Any biopsies will be performed by the health care provider as a standard of care procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female all age groups
* Ability to understand and carry out subject instructions

Exclusion Criteria:

* Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be selected from University of California Irvine Medical Clinic
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-04; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
high-resolution images of skin | up to 12 months
  The complementary imaging modalities (MPM, MI) will provide insights into a better understanding of the relationship between microscopic and macroscopic properties of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No